CLINICAL TRIAL: NCT03002038
Title: Comparison of Annual Relapse Rate, Expanded Disability Status Scale, and Side Effects Between Azathioprine and Rituximab in Patients With Neuromyelitis Optica Spectrum Disorders
Brief Title: Comparison of Clinical Effects of Azathioprine and Rituximab NMO-SD Patients
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Isfahan University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Vahid Shaygannejad, Associate Professor of Neurology, Isfahan University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 395275
Record Dates: First submitted 2016-12-21; First posted 2016-12-23 (Estimated); Results first posted 2020-09-30 (Actual); Last update posted 2020-09-30 (Actual); Status verified 2020-09

CONDITIONS: Neuromyelitis Optica Spectrum Disorder
Keywords: neuromyelitis optica spectrum disorder; azathioprine; rituximab; clinical trial; annual relapse rate; expanded disability status scale
MeSH Terms: conditions — Neuromyelitis Optica | interventions — Azathioprine; Rituximab; Reditux

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Azathioprine (Experimental): Patients in this group will receive 50 mg of azathioprine, two times each day and gradually increased to maximum dose of 3 g daily with the aim of lymphocytes count less than 1500.
  Interventions: Drug: Azathioprine
- Rituximab (Experimental): Patients in this group will receive 1g of Rituximab in 500 cc normal saline serum through intravenous infusion with two weeks intervals (as one course) and each course of treatment is repeated every 6 months.
  Interventions: Drug: Rituximab

INTERVENTIONS:
Drug: Azathioprine — Patients are started with Azathioprine 50 mg tablets, taken orally twice a day. The medication dose is increased gradually with the aim of lymphocytes count bellow 1500 and to the maximum dose of 3 g Azathioprine per day. Cell blood count is checked once a week in the first month of treatment, once every two weeks in the second month of treatment, and monthly in the third month of treatment to make decision about medication dose.
  Other Names: Azathioprine Mehrdaru®
  Arms: Azathioprine
Drug: Rituximab — Patients will receive 1 g of Rituximab (two vials of RediTux 500 mg/50 ml) in 500 cc normal saline serum through intravenous infusion and this will be repeated two weeks later. This cycle will be repeated every 6 months.
  Other Names: RediTux®
  Arms: Rituximab

SUMMARY:
The purpose of this study is to compare annual relapse rate, expanded disability status scale, and side effects of azathioprine and rituximab in patients with neuromyelitis optica spectrum disorder during a one year follow up through a randomized clinical trial.

DETAILED DESCRIPTION:
Neuromyelitis Optica Spectrum Disorder (NMO-SD) is a recurrent inflammatory demyelinating disease affecting the central nervous system. The disease is clinically recognized by optic neuritis and transverse myelitis and is associated with high risk of mortality. Each attack worsens patients' disability. This means that after 5 years of the disease onset, half of patients need to use wheelchair and approximately 50% of them become blind.

Considering that the disease can be disabling for patients, the maintenance treatment should be applied in addition to treatment of acute attacks, in order to prevent future recurrences. Acute attacks are usually treated with high doses of intravenous corticosteroids. Plasmapheresis is also used when patients fail to response to corticosteroids. B lymphocyte inhibitors are used as the maintenance therapy in these patients. First line therapeutic medications include azathioprine and rituximab which are being recommended for long term therapy and second line medications include methotrexate and mycophenolate mofetil.

Azathioprine is an immune-modulatory agent which is available in the oral form and don't require hospitalization to be administered, however, because of side effects such as bone marrow suppression and hepatotoxicity, periodic check of blood cells and liver enzymes are needed. Rituximab is a cluster of differentiation antigen 20 inhibitor which leads to decreased B lymphocytes and antibody in patients. This medication is only available in the injectable form and needs hospitalization to be administered. Close monitory is needed during the administration considering severe side effects such as allergic reactions and respiratory distress. However, laboratory tests are not needed in patients taking rituximab although it is more expensive than azathioprine. No clinical trial has been performed previously to compare clinical efficacy of these two drugs in NMO-SD patients. Therefore, we aimed to compare their efficacy through a randomized clinical trial.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of neuromyelitis optica spectrum disorder based on the recent guidelines in 2015
* Expanded disability status scale between 0 and 7
* Age between 18 and 50 years old

Exclusion Criteria:

* Pregnancy or lactation during the study
* Deciding to leave the study by patient
* Lack of consent to enter the study
* Lack of cooperation for follow up
* Severe side effect of the medication
* Treatment with other immunosuppressant medications (including but not limited to cyclophosphamide, mycophenolate mofetil, methotrexate, others) within two months before intervention
* Taking any other immunosuppressant or other type of medication (including herbal drugs) without permission of the physician during the study.
* Presence of other autoimmune disease (including but not limited to Behcet disease, systemic lupus erythematosus, rheumatoid arthritis, and others)
* Presence of liver disorders
* Presence of hematologic disorders
* Presence of heart failure
* Receipt of a live vaccine within 4 weeks prior to intervention
* Previous treatment with Azathioporine or Rituximab
* History of HIV, hepatitis B, or hepatitis C
* Ongoing daily steroid use
* History of severe allergic or anaphylactic reaction to monoclonal antibodies

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 86 (Actual)
Dates: Start 2015-09; Primary Completion 2016-11 (Actual); Study Completion 2016-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Vahid Shaygannejad, M.D., Study Chair — Department of Neurology, School of Medicine, Isfahan University of Medical Sciences
Locations (1):
- Kashani Hospital, Isfahan, Iran

IPD SHARING:
Plan to Share IPD: Undecided
We may share the individual participant data (anonymously) on request of the journal publishing the study report.

REFERENCES:
- [Background] Sato DK, Lana-Peixoto MA, Fujihara K, de Seze J. Clinical spectrum and treatment of neuromyelitis optica spectrum disorders: evolution and current status. Brain Pathol. 2013 Nov;23(6):647-60. doi: 10.1111/bpa.12087. PMID 24118482
- [Background] Morrow MJ, Wingerchuk D. Neuromyelitis optica. J Neuroophthalmol. 2012 Jun;32(2):154-66. doi: 10.1097/WNO.0b013e31825662f1. PMID 22617743
- [Background] Costanzi C, Matiello M, Lucchinetti CF, Weinshenker BG, Pittock SJ, Mandrekar J, Thapa P, McKeon A. Azathioprine: tolerability, efficacy, and predictors of benefit in neuromyelitis optica. Neurology. 2011 Aug 16;77(7):659-66. doi: 10.1212/WNL.0b013e31822a2780. Epub 2011 Aug 3. PMID 21813788
- [Background] Trebst C, Jarius S, Berthele A, Paul F, Schippling S, Wildemann B, Borisow N, Kleiter I, Aktas O, Kumpfel T; Neuromyelitis Optica Study Group (NEMOS). Update on the diagnosis and treatment of neuromyelitis optica: recommendations of the Neuromyelitis Optica Study Group (NEMOS). J Neurol. 2014 Jan;261(1):1-16. doi: 10.1007/s00415-013-7169-7. Epub 2013 Nov 23. PMID 24272588
- [Background] Kim SH, Huh SY, Lee SJ, Joung A, Kim HJ. A 5-year follow-up of rituximab treatment in patients with neuromyelitis optica spectrum disorder. JAMA Neurol. 2013 Sep 1;70(9):1110-7. doi: 10.1001/jamaneurol.2013.3071. PMID 23897062
- [Background] Katz Sand I. Neuromyelitis Optica Spectrum Disorders. Continuum (Minneap Minn). 2016 Jun;22(3):864-96. doi: 10.1212/CON.0000000000000337. PMID 27261687
- [Derived] Nikoo Z, Badihian S, Shaygannejad V, Asgari N, Ashtari F. Comparison of the efficacy of azathioprine and rituximab in neuromyelitis optica spectrum disorder: a randomized clinical trial. J Neurol. 2017 Sep;264(9):2003-2009. doi: 10.1007/s00415-017-8590-0. Epub 2017 Aug 22. PMID 28831548

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Azathioprine | Rituximab
Started | 46 | 40
Completed | 35 | 33
Not Completed | 11 | 7
Not completed — Adverse Event | 3 | 1
Not completed — Withdrawal by Subject | 8 | 4
Not completed — Immigration to another region | 0 | 2

BASELINE CHARACTERISTICS:
Population: Intention to treat analysis
Groups:
- Total: Total of all reporting groups
Arm/Group | Azathioprine | Rituximab | Total
Number analyzed (Participants) | 46 | 40 | 86
Age, Continuous [Mean (Standard Deviation); unit: years] | 32.11 (9.36) | 34.33 (5.86) | 33.14 (7.32)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 38 | 34 | 72
  Male | 8 | 6 | 14
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Iran | 46 | 40 | 86
Expanded disability status scale [Mean (Standard Deviation); unit: units on a scale] — Expanded disability status scale (EDSS) is a measure of disability for patients. The score ranges from 0-10, with 0 showing normal neurological exam and 10 showing death due to the disabling disease. Thus, higher scores represent more profound levels of disability. Population: Per reviewer's comment and to provide consistent results, we changed the baseline info for EDSS to per protocol analysis rather than intended to treat analysis. That's why the numbers decreased in each group.
  units on a scale
    number analyzed (Participants) | 35 | 33 | 68
    (all) | 2.40 (1.24) | 3.55 (1.95) | 2.96 (1.52)
Annualized relapse rate [Mean (Standard Deviation); unit: numbers of relapses] | 1.02 (0.39) | 1.30 (0.65) | 1.15 (0.51)
Positive AQP4-IgG [Count of Participants; unit: Participants] | 25 | 17 | 42

OUTCOME MEASURES:

1. Primary Outcome: Annual Relapse Rate
Description: annual relapse rate will be measured in the baseline (according to patients' history in the last year) and after 12 months of intervention.
Time Frame: one year
Population: Per protocol analysis
Measure: Mean (Standard Deviation); unit: Number of relapses
Arm/Group | Azathioprine | Rituximab
Number analyzed (Participants) | 35 | 33
Number of relapses
  Baseline | 1 (0.38) | 1.30 (0.68)
  Outcome | 0.51 (0.55) | 0.21 (0.42)

2. Secondary Outcome: Expanded Disability Status Scale
Description: expanded disability status scale will be measured in the baseline and after 12 months of intervention.
  Expanded disability status scale (EDSS) is a measure of disability for patients. The score ranges from 0-10, with 0 showing normal neurological exam and 10 showing death due to the disabling disease. Thus, higher scores represent more profound levels of disability.
Time Frame: one year
Population: Per protocol analysis
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Azathioprine | Rituximab
Number analyzed (Participants) | 35 | 33
score on a scale
  Baseline | 2.40 (1.24) | 3.55 (1.95)
  Outcome | 1.95 (1.13) | 2.56 (1.99)

3. Other Pre Specified Outcome: Number of Participants With Adverse Drug Reactions
Description: adverse drug reactions will be observed closely and reported during the intervention. We will compare the number of adverse drug reactions in two groups. Also, adverse drug reactions will be described by details in each group.
Time Frame: one year
Population: intention to treat analysis
Measure: Count of Participants; unit: Participants
Arm/Group | Azathioprine | Rituximab
Number analyzed (Participants) | 46 | 40
Participants | 3 | 4

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Azathioprine | Rituximab
All-Cause Mortality (participants affected / at risk) | 0/46 | 0/40
Serious Adverse Events (participants affected / at risk) | 1/46 | 1/40
Other Adverse Events (participants affected / at risk) | 2/46 | 3/40
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Azathioprine (N=46) | Rituximab (N=40)
Impaired liver function test (Hepatobiliary disorders) | 1 (1) | 0 (0)
Severe allergic reaction (Immune system disorders) | 0 (0) | 1 (1) — Allergic reaction to rituximab injection
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Azathioprine (N=46) | Rituximab (N=40)
Mild/moderate allergic reactions (Immune system disorders) | 0 (0) | 3 (3)
Gastrointestinal intolerance (Gastrointestinal disorders) | 2 (2) | 0 (0)

LIMITATIONS AND CAVEATS:
lack of blinding, uneven assignment of patients to treatment groups, lack of compliance measures, and short follow-up duration

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes